CLINICAL TRIAL: NCT04338529
Title: Alendronate in an Weekly Effervescent Tablet Formulation for Preservation of Bone Mass After Denosumab Discontinuation in Postmenopausal Women with Low Bone Mass. an Observational Study (Binosto After Denosumab - the BAD Study)
Brief Title: Alendronate in an Weekly Effervescent Tablet Formulation Following Denosumab Discontinuation
Acronym: BAD
Status: Completed | Type: Observational
Sponsor: 251 Hellenic Air Force & VA General Hospital (Other)
Collaborators: Laikο General Hospital, Athens (Other); 424 General Military Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: F076/AD1704/S606/18-2-2020; 2550/14-2-20 (Other: LAIKO Hospital)
Record Dates: First submitted 2020-04-04; First posted 2020-04-08 (Actual); Last update posted 2024-12-02 (Actual); Status verified 2024-11

CONDITIONS: Postmenopausal Osteoporosis
Keywords: Denosumab; Alendronate; osteoporosis; discontinuation of treatment
MeSH Terms: conditions — Osteoporosis, Postmenopausal; Osteoporosis | interventions — Alendronate; Calcium Carbonate; Cholecalciferol

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Morning (8-9 am) fasting blood samples will be obtained at baseline and at 3, 6, 9 and 12 months. Blood samples will be centrifuged immediately and serum will be separated and stored at -80 ºC; 24hours urine specimens will be collected at 6 and 12 months.
  All study parameters will be measured in one batch at the end of the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Group Alendronate 6m: Postmenopausal Caucasian women who were treated with denosumab and became osteopenic (BMD T-score of > -2.5 at the LS and the non-dominant FN) and were assigned from their treating physician to receive treatment with alendronate in an effervescent tablet formulation for 6 months and then followed for another 6 months without medication. In case serum P1NP levels are > 35μg/L and/or serum CTX levels are > 280 ng/L at 9 months (3 months following alendronate discontinuation) the patients would be strongly advised to restart alendronate treatment.
  Interventions: Drug: Binosto 70Mg Effervescent Tablet
- Group Alendronate 12m: Postmenopausal Caucasian women who were treated with denosumab and became osteopenic (BMD T-score of > -2.5 at the LS and the non-dominant FN) and were assigned from their treating physician to receive treatment with alendronate in an effervescent tablet formulation for 12 months.
  Interventions: Drug: Binosto 70Mg Effervescent Tablet

INTERVENTIONS:
Drug: Binosto 70Mg Effervescent Tablet — As discussed in group descriptions
  Other Names: calcium carbonate 1000 mg/d and cholecalciferol 800 IU/d

SUMMARY:
Discontinuation of denosumab results in a rebound response of bone turnover markers, which rise above baseline at 3 months and remain elevated until reaching again baseline levels approximately 30 months after the last dose. Bone mineral density (BMD) gains are also lost and BMD values reach original baseline values after 1-2 years off-treatment.For the above reasons, current literature recommends that patients who discontinue denosumab should continue to receive either intravenous (iv) or oral (peros) bisphosphonate therapy for some time. The study aims to investigate changes in the BMD of the lumbar spine 12 months after transitioning from denosumab to oral alendronate 70 mg in a weekly effervescent tablet formulation

DETAILED DESCRIPTION:
Denosumab, a monoclonal antibody against the receptor activator of nuclear factor κ-Β ligand (RANKL), is a potent antiresorptive agent commonly prescribed in patients with postmenopausal osteoporosis. Discontinuation of denosumab results in a rebound response of bone turnover markers, which rise above baseline at 3 months and remain elevated until reaching again baseline levels approximately 30 months after the last dose. Bone mineral density (BMD) gains are also lost and BMD values reach original baseline values after 1-2 years off-treatment, in contrast to bisphosphonates, which remain within the skeleton acting for several months or even years after discontinuation while preserving most of the BMD gains achieved despite the cessation of treatment.

For the above reasons, current literature recommends that patients who discontinue denosumab should continue to receive either intravenous (iv) or oral (peros) bisphosphonate therapy for some time. Due to lack of specifically designed studies, the period of treatment with bisphosphonates after denosumab discontinuation has been arbitrarily proposed to be 1 to 2 years. Preservation of BMD gains after denosumab discontinuation has so far been demonstrated: (a) with one year of alendronate treatment, in a study designed to investigate patients' compliance to treatment, and b) with a single dose of zolendronate 5mg iv in a recent study specifically designed to address this question in which BMD levels remained stable for the next two years.

Preventing bone loss, and the reported high risk of multiple vertebral fractures after discontinuation of denosumab treatment, is a clinical issue of critical importance raising serious concerns to the international scientific community and needs to be addressed. Clinical studies specifically designed to investigate both the efficacy of various bisphosphonates and the optimal duration of their administration in order to avoid the reported adverse effects of denosumab discontinuation are currently lacking.

This study aims to investigate changes in the BMD of the lumbar spine (LS) and femoral neck (FN) 12 months after transitioning from denosumab to oral alendronate 70 mg in a weekly effervescent tablet formulation. Alendronate will be given either for 6 or 12 months following Denosumab discontinuation

ELIGIBILITY:
Inclusion Criteria:

i) osteopenic postmenopausal Caucasian women following Dmab treatment ii) assignment to treatment with alendronate in an effervescent tablet formulation following Dmab discontinuation

Exclusion Criteria:

i) secondary osteoporosis; ii) diseases that could affect bone metabolism iii) medications that could affect bone metabolism iv) chronic kidney disease (stage >3b) and/or liver failure v) neoplastic disease vi) hypersensitivity to alendronate or to any of the excipients vii) abnormalities of the esophagus and other factors which delay esophageal emptying such as stricture or achalasia viii) inability to stand or sit upright for at least 30 minutes ix) hypocalcaemia x) confirmed esophagitis

Max Age: 90 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study will include postmenopausal Caucasian women who were treated with denosumab and became osteopenic (BMD T-score of > -2.5 at the LS and the non-dominant FN) and were assigned from their treating physician to receive treatment with alendronate in an effervescent tablet formulation for either 6 months (Group 6, n=46) and then followed for another 6 months without medication, or 12 months of continuous treatment with alendronate (Group 12, n=46). As this is an observational study, patients could be either referred from their treating physicians or could be actually followed by the investigators themselves in case the investigator is the treating physician
Sampling Method: Non-Probability Sample
Enrollment: 92 (Actual)
Dates: Start 2020-04-01 (Actual); Primary Completion 2024-09-25 (Actual); Study Completion 2024-11-01 (Actual)

PRIMARY OUTCOMES:
Bone Mineral Density LS | 12 months
  Changes in the BMD of the lumbar spine 12 months after transitioning from denosumab to oral alendronate 70 mg in a weekly effervescent tablet formulation.

SECONDARY OUTCOMES:
Bone Mineral Density FN | 12 months
  Changes in the BMD of the femoral neck (FN) of the non-dominant hip 12 months after transitioning from denosumab to oral alendronate 70 mg in a weekly effervescent tablet formulation
Serum levels of bone turnover markers (BTMs): P1NP, CTX and TRAP5b | 12 months
  Changes in BTMs 12 months after transitioning from denosumab to oral alendronate 70mg in a weekly effervescent tablet formulation.
Comparison of Bone Mineral Density LS | 12 months
  Comparison of changes in the BMD of the LS after transitioning from denosumab to 12 months versus 6 months of treatment with oral alendronate 70 mg in a weekly effervescent tablet formulation.
Comparison of Bone Mineral Density FN | 12 months
  Comparison of changes in the BMD of the FN of the non-dominant hip after transitioning from denosumab to 12 months versus 6 months of treatment with oral alendronate 70mg in a weekly effervescent tablet formulation.
Comparison of changes in: the serum levels of bone turnover markers (BTMs) P1NP, CTX and TRAP5b; the 24-hours urine levels of calcium | 12 months
  Comparison of changes in the levels of serum BTMs and 24hours urine calcium after 12 months versus 6 months treatment with oral alendronate 70mg in a weekly effervescent tablet formulation in patients previously treated with denosumab

CONTACTS AND LOCATIONS:
Overall Officials: Maria Yavropoulou, MD, PhD, Study Chair — LAIKO General Hospital, Athens, Greece; Polyzois Makras, MD, PhD, Principal Investigator — 251 Hellenic Airforce Gen. Hospital, Athens, Greece; Athanasios D Anastasilakis, MD, PhD, Study Director — 424 Gen. Military Hospital Thessaloniki, Greece
Locations (1):
- 251 Hellenic Air Force & VA General Hospital, Athens, Attica, Greece

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cummings SR, San Martin J, McClung MR, Siris ES, Eastell R, Reid IR, Delmas P, Zoog HB, Austin M, Wang A, Kutilek S, Adami S, Zanchetta J, Libanati C, Siddhanti S, Christiansen C; FREEDOM Trial. Denosumab for prevention of fractures in postmenopausal women with osteoporosis. N Engl J Med. 2009 Aug 20;361(8):756-65. doi: 10.1056/NEJMoa0809493. Epub 2009 Aug 11. PMID 19671655
- [Background] Miller PD, Bolognese MA, Lewiecki EM, McClung MR, Ding B, Austin M, Liu Y, San Martin J. Effect of denosumab on bone density and turnover in postmenopausal women with low bone mass after long-term continued, discontinued, and restarting of therapy: a randomized blinded phase 2 clinical trial. Bone. 2008 Aug;43(2):222-229. doi: 10.1016/j.bone.2008.04.007. Epub 2008 Apr 26. PMID 18539106
- [Background] Bone HG, Bolognese MA, Yuen CK, Kendler DL, Miller PD, Yang YC, Grazette L, San Martin J, Gallagher JC. Effects of denosumab treatment and discontinuation on bone mineral density and bone turnover markers in postmenopausal women with low bone mass. J Clin Endocrinol Metab. 2011 Apr;96(4):972-80. doi: 10.1210/jc.2010-1502. Epub 2011 Feb 2. PMID 21289258
- [Background] McClung MR, Wagman RB, Miller PD, Wang A, Lewiecki EM. Observations following discontinuation of long-term denosumab therapy. Osteoporos Int. 2017 May;28(5):1723-1732. doi: 10.1007/s00198-017-3919-1. Epub 2017 Jan 31. PMID 28144701
- [Background] Anastasilakis AD, Polyzos SA, Makras P, Aubry-Rozier B, Kaouri S, Lamy O. Clinical Features of 24 Patients With Rebound-Associated Vertebral Fractures After Denosumab Discontinuation: Systematic Review and Additional Cases. J Bone Miner Res. 2017 Jun;32(6):1291-1296. doi: 10.1002/jbmr.3110. Epub 2017 Mar 13. PMID 28240371
- [Background] Cummings SR, Ferrari S, Eastell R, Gilchrist N, Jensen JB, McClung M, Roux C, Torring O, Valter I, Wang AT, Brown JP. Vertebral Fractures After Discontinuation of Denosumab: A Post Hoc Analysis of the Randomized Placebo-Controlled FREEDOM Trial and Its Extension. J Bone Miner Res. 2018 Feb;33(2):190-198. doi: 10.1002/jbmr.3337. Epub 2017 Nov 22. PMID 29105841
- [Background] Black DM, Bauer DC, Schwartz AV, Cummings SR, Rosen CJ. Continuing bisphosphonate treatment for osteoporosis--for whom and for how long? N Engl J Med. 2012 May 31;366(22):2051-3. doi: 10.1056/NEJMp1202623. Epub 2012 May 9. No abstract available. PMID 22571169
- [Background] Anastasilakis AD, Polyzos SA, Makras P. THERAPY OF ENDOCRINE DISEASE: Denosumab vs bisphosphonates for the treatment of postmenopausal osteoporosis. Eur J Endocrinol. 2018 Jul;179(1):R31-R45. doi: 10.1530/EJE-18-0056. Epub 2018 Apr 24. PMID 29691303
- [Background] Tsourdi E, Langdahl B, Cohen-Solal M, Aubry-Rozier B, Eriksen EF, Guanabens N, Obermayer-Pietsch B, Ralston SH, Eastell R, Zillikens MC. Discontinuation of Denosumab therapy for osteoporosis: A systematic review and position statement by ECTS. Bone. 2017 Dec;105:11-17. doi: 10.1016/j.bone.2017.08.003. Epub 2017 Aug 5. PMID 28789921
- [Background] Freemantle N, Satram-Hoang S, Tang ET, Kaur P, Macarios D, Siddhanti S, Borenstein J, Kendler DL; DAPS Investigators. Final results of the DAPS (Denosumab Adherence Preference Satisfaction) study: a 24-month, randomized, crossover comparison with alendronate in postmenopausal women. Osteoporos Int. 2012 Jan;23(1):317-26. doi: 10.1007/s00198-011-1780-1. Epub 2011 Sep 17. PMID 21927922
- [Background] Anastasilakis AD, Papapoulos SE, Polyzos SA, Appelman-Dijkstra NM, Makras P. Zoledronate for the Prevention of Bone Loss in Women Discontinuing Denosumab Treatment. A Prospective 2-Year Clinical Trial. J Bone Miner Res. 2019 Dec;34(12):2220-2228. doi: 10.1002/jbmr.3853. Epub 2019 Oct 14. PMID 31433518